CLINICAL TRIAL: NCT03147443
Title: The Study on the Effects of Traditional Chinese Medicine Through a Series of N-of-1 Trials Based on the Mathematical Model of "Carryover Effect"
Brief Title: Evaluating the Effects of Traditional Chinese Medicine by N-of-1 Trials
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, haiyinhuang, chief physician, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: haiyinhuang
Record Dates: First submitted 2017-05-03; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Bronchiectasis; Quality of Life; Traditional Chinese Medicine; Sputum; Symptoms; Individuality
Keywords: traditional Chinese medicine; Drugs, Chinese Herbal; N-of-1 trials; sputum; symptoms; individualized treatment; stable bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, crossover comparisons of individualized herbal decoction with control decoction within individual patients. Each n-of-1 trial has 3 pairs of treatment periods. The duration of each treatment period will be 4 weeks.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Placebo is made by dextrin, bitter agent, edible pigment etc and added 5% test drug. The test drug and control drug have no differences in dosage form, appearance, color, specification, label, and so forth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized Decoction (Experimental): It is the highly individualized treatment of traditional Chinese medicine,the modification of Bronchiectasis Stabilization Decoction(Radix Lithospermi 15 g, Rhizoma Fagopyri Cymosi 30 g, Radix Ophiopogonis 15 g, Poria cocos 15 g, Radix Astragali 20 g, Rhizoma Bletillae 10 g, Platycodon grandiflorum 10 g, and Semen Coicis 30 g) based on syndrome differentiation. For example,for patients with qi and yin deficiency syndrome, we added Radix Adenophorae, and Radix Rehmanniae Recens. Besides, the herbs in a prescription could be changed according to different symptoms of individual patients.
  The Chinese herbal decoction is taken by one decoction a day and divided into 2 doses, for 3 weeks in each observation period.
  Interventions: Drug: Individualized Decoction; Drug: placebo
- placebo (Placebo Comparator): Placebo is made by dextrin, bitter agent, edible pigment etc and added 5% test drug. The placebo and test drug have no differences in dosage form, appearance, color, specification, label, and so forth.
  The placebo is taken by one decoction a day and divided into 2 doses, for 3 weeks in each observation period.
  Interventions: Drug: Individualized Decoction; Drug: placebo
- Tested drug minus heat-clearing herbs (Active Comparator): It is the decoction of the Individualized Syndrome Differentiation Decoction(tested drug) minus heat-clearing herbs. For example, heat-clearing herbs such as Scutellaria baicalensis or Herba Violae will be removed from the Syndrome Differentiation Decoction.
  This control Chinese herbal decoction is taken by one decoction a day and divided into 2 doses, for 3 weeks in each observation period.
  Interventions: Drug: Individualized Decoction; Drug: Tested drug minus heat-clearing herbs

INTERVENTIONS:
Drug: Individualized Decoction — Applied in the Tested Drug Observation Period. It is the highly individualized treatment of traditional Chinese medicine,the modification of Bronchiectasis Stabilization Decoction(Radix Lithospermi 15 g, Rhizoma Fagopyri Cymosi 30 g, Radix Ophiopogonis 15 g, Poria cocos 15 g, Radix Astragali 20 g, Rhizoma Bletillae 10 g, Platycodon grandiflorum 10 g, and Semen Coicis 30 g) based on syndrome differentiation. For example,for patients with qi and yin deficiency syndrome, we added Radix Adenophorae, and Radix Rehmanniae Recens. Besides, the herbs in a prescription could be changed according to different symptoms of individual patients.
Drug: placebo — Applied in the placebo Observation Period. Placebo is made by dextrin, bitter agent, edible pigment etc and added 5% test drug. The test drug and control drug have no differences in dosage form, appearance, color, specification, label, and so forth.
  Arms: Individualized Decoction; placebo
Drug: Tested drug minus heat-clearing herbs — It is the decoction of the Syndrome Differentiation Decoction(tested drug) minus heat-clearing herbs. For example, heat-clearing herbs such as Scutellaria baicalensis or Herba Violae will be removed from the Syndrome Differentiation Decoction.
  Arms: Tested drug minus heat-clearing herbs

SUMMARY:
Treatment based on syndrome differentiation is the essence of traditional Chinese Medicine(TCM) and forms the individualized treatment. N-of-1 trials may be a good clinical effect evaluation method for the individualized treatment of TCM. This study aims to compare: (1) the efficacy of syndrome differentiation(individualized decoction) with placebo, (2)the efficacy of syndrome differentiation(individualized decoction) with the same prescription minus heat-clearing Chinese herbs, for patients with stable bronchiectasis through N-of-1 trials.

DETAILED DESCRIPTION:
Traditional Chinese medicine is one of the important part of complementary and alternative medicine in the world, and it plays increasingly important role in the international medical practice. Treatment based on syndrome differentiation is the essence of traditional Chinese Medicine (TCM) and forms the individualized treatment. However, this individualized TCM intervention often makes it difficult for population-based RCTs to carry out a standard form. N-of-1 trials may be a good clinical effect evaluation method for the individualized treatment of TCM.

The key hypothesis of this study is that: (1) the efficacy of syndrome differentiation(individualized decoction) will be better than placebo in patients with stable bronchiectasis through N-of-1 trials. (2) the efficacy of syndrome differentiation(individualized decoction) will be better than the same prescription minus heat-clearing Chinese herbs in patients with stable bronchiectasis through N-of-1 trials. The difference of efficacy may be various according to the individual severity of phlegm-heat.

In this study, We will conduct a single center N-of-1 trials in 36 patients with stable bronchiectasis without hemoptysis and respiratory failure. These N-of-1 trials will be randomized, double-blind, crossover comparisons of individualized herbal decoction with control decoction within individual patients. Each n-of-1 trial has 3 pairs of treatment periods. The duration of each treatment period will be 4 weeks. We will compare :(1) the efficacy of syndrome differentiation(individualized decoction) with placebo, (2) the efficacy of syndrome differentiation(individualized decoction) with the same prescription minus heat-clearing Chinese herbs, in patients with stable bronchiectasis through N-of-1 trials. The primary outcome is patient self-reported symptoms(such as cough, expectoration, shortness of breath, chest pain, and fatigue) scores on a 7 point visual analogue scale. Secondary outcomes are 24-hour sputum volume and CAT（The COPD Assessment Test） scores. We use paired t test for single case. Mixed effects model taking account of "Carryover Effects" and meta-analysis will be used for a series of N-of-1 trials as a group.

ELIGIBILITY:
Inclusion Criteria:

* the diagnostic criteria based on the consensus of Chinese experts and the guidelines for noncystic fibrosis bronchiectasis issued by the British Thoracic Society in 2010;
* male or female, aged 18-70 years;
* being in the stable stage, and no acute exacerbation of bronchiectasis within the past three weeks;
* frequency of acute exacerbation of bronchiectasis ≤ 3 times every year;
* signed informed consent for participation.

Exclusion Criteria:

* having developed respiratory failure with estimated survival time less than one year;
* having hemoptysis as a comorbidity;
* having complications by active tuberculosis;
* being pregnant or with severe heart, liver,and kidney dysfunctions;
* participating in other pharmacological clinical trials within the past 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Self-Rated Symptom Score | 4 weeks
  Patients rated the severity of the symptoms (such as cough, expectoration, shortness of breath, chest pain, and fatigue) on a 7 point visual analogue scales. The higher the score, the more severe the symptom.

SECONDARY OUTCOMES:
24 h Sputum Volume | 4 weeks
  We measured the 24h sputum volume at the beginning and the end of each treatment period of the trial. To ensure the accuracy of the measurement, we asked the patients to spit sputum into a collector with scales from 8:00 am to the next 8:00 am. We used the mean value of the sputum volume for 3 consecutive days as the outcome.

OTHER OUTCOMES:
COPD Assessment Test | 4 weeks
  COPD Assessment Test questionnaire is composed of 8 items. Each item has a score ranging from 0 to 5, thereby making the total score range from 0 to 40. Score of 0 represents the best quality of life and 40 does the worst.

CONTACTS AND LOCATIONS:
Locations (1):
- Yueyang Hospital of Integrated Traditional Chinese and Western Medicine,Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang H, Yang P, Xue J, Tang J, Ding L, Ma Y, Wang J, Guyatt GH, Vanniyasingam T, Zhang Y. Evaluating the Individualized Treatment of Traditional Chinese Medicine: A Pilot Study of N-of-1 Trials. Evid Based Complement Alternat Med. 2014;2014:148730. doi: 10.1155/2014/148730. Epub 2014 Nov 11. PMID 25477988
- [Background] Lee BY, Lee S, Lee JS, Song JW, Lee SD, Jang SH, Jung KS, Hwang YI, Oh YM. Validity and Reliability of CAT and Dyspnea-12 in Bronchiectasis and Tuberculous Destroyed Lung. Tuberc Respir Dis (Seoul). 2012 Jun;72(6):467-74. doi: 10.4046/trd.2012.72.6.467. Epub 2012 Jun 29. PMID 23101012
- [Derived] Zi S, Huang H, Yang P, Xu M, Wu Y, Wang Z, Ge F, Chen X. Evaluating the Effects of Heat-Clearing Traditional Chinese Medicine in Stable Bronchiectasis by a Series of N-of-1 Trials. Evid Based Complement Alternat Med. 2022 Jan 17;2022:6690638. doi: 10.1155/2022/6690638. eCollection 2022. PMID 35087595